CLINICAL TRIAL: NCT05514223
Title: MeaSuring Free radIcals With Diamond magnetometrRy In hUman Single Sperm Cells Related to Microbiota and Lifestyle Factors
Brief Title: Measuring Free Radicals in Human Sperm Cells Related to Microbiota and Lifestyle Factors
Acronym: SIRIUS
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 202100341
Record Dates: First submitted 2022-02-15; First posted 2022-08-24 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Infertility, Male; Infertility
Keywords: Free radicals; Reactive oxygen species; Microbiota; Diet; Dietary patterns; Fertility; Semen analysis; Fertility clinics; Diamond magnetometry; Lifestyle; Semen; Oxidative stress; Food frequency questionnaire
MeSH Terms: conditions — Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Semen (whole ejaculate) and blood plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Males of couples seeking fertility treatment: The study population will consist of males of couples that visit the Center reproductive Medicine of the UMCG where a semen analysis is planned for clinical purposes.
  Interventions: Other: Biomaterial collection for observational purpose

INTERVENTIONS:
Other: Biomaterial collection for observational purpose — The semen will be collected to measure the free radical concentration in seminal plasma and sperm together with the diversity of microbiota. Both males with a normal semen analysis (SA) and abnormal SA according to the WHO guidelines (2010) will be included. Blood plasma will be collected to measure systemic radical concentration and all outcomes will be related to lifestyle factors and food intake acquired through hospital charts and routinely conducted questionnaires together with a food frequency Questionnaire (FFQ).

SUMMARY:
The cause of infertility can be due to a female factor or a male factor. In case of a male factor, it is often due to poor semen quality. However, the cause of poor quality is often unknown. In previous research, infertility problems in men were related to chemical processes in metabolism causing the formation of free radicals. Free radicals are physiological by-products of our body mechanisms. Free radicals are very reactive and can therefore react with a lot of molecules of cells within our body and cause damage. A balance between free radicals, which are also needed for physiological processes in the body, and antioxidants, which defuses the reactive free radicals, is most desirable. However, as stated in literature, there are a lot of factors that can influence extra free radical production, which causes overloading of the system, resulting in damage on cellular level. Free radicals in semen plasma and on the sperm cell could play a role in male infertility. Nonetheless, free radicals are not used as diagnostic markers due to the lack of detection systems, as free radicals are very short-lived. This study aims to introduce a new technique, called diamond magnetometry, to measure free radicals directly on the sperm cell and in serum. Diamond magnetometry involves very small diamond particles as magnetic sensors that engage a reaction with the free radicals on the sperm cell, causing signals that can be measured. To compare local free radical production with systemic free radical production, other diagnostic biomarkers are also measured in serum.

It is hypothesized that the composition of seminal microbiome could influence the free radical concentration. Therefore, this study also aims to explore the microbiota composition and see if this has an influence in semen quality and free radical production. At last, this study also want to correlate standard semen parameters (defined by the World Health Organisation), lifestyle factors and food intake, to detect a role for lifestyle in the production of free radicals.

DETAILED DESCRIPTION:
To date, 15% of couples experience issues with fertility and in 40-50% of the cases it is thought to be due to fertility issues in men. Reactive oxygen species (ROS) and especially free radicals (the most reactive ones) play a key role in sperm capacitation and fertilisation. They are also believed to be a major contributor to male infertility. The free radical theory of infertility states that damage by free radicals is the main cause of infertility in males. However, they are difficult to measure due to their short lifetime and high reactivity.

Despite the relevance of free radicals, they are not used as diagnostic biomarkers nor as target for therapeutics since it is currently unknown where and when the free radicals are generated exactly, due to the insufficiency of the currently available techniques. Therefore, a new technique will be utilized called diamond magnetometry which allows nanoscale magnetic resonance measurements. This quantum sensing technique is uniquely sensitive and allows real-time single cell measurements with sub-cellular resolution. Unlike most other techniques this method is specific for free radicals. A first proof of principle experiment has been published in yeast cells and we have preliminary data which proofs that we can measure free radical generation in boar sperm. The concentration of free radicals will be related to standard semen-parameters according to the WHO guidelines, lifestyle factors and food intake and related with microbiota in semen plasma to explore possible correlations. Microbiota have been suggested to play a role in the context of reproduction. While several studies have been carried out focusing on the female reproductive system, less is known about male microbiota and its influence on fertility. In the past it was thought that the presence of bacteria in the semen was an indicator of infection. The next generation genetic-based approach has revealed that the human semen is not sterile and appear to host a specific microbiota. Alterations of the diversity of seminal microbiota or the abundance of specific bacteria have been associated with an altered morphology and motility of sperm cells. Nevertheless, the molecular processes through which bacteria are able to alter semen quality are unknown. Possible mechanisms may involve free radical damaging or alteration of other molecules (e.g. lipids peroxidation, DNA fragmentation) which may result in loss of fertilisation capability. Therefore, it is hypothesized that free radical generation is correlated to the diversity of microbiota and can be related to the semen-parameters defined by the WHO guidelines.

The primary objective of this study is to measure real-time free radicals in human single sperm cells using diamond magnetometry. This is correlated to the seminal microbiota composition to investigate the influence of the composition in free radical generation, and therefore a possible mechanism of microorganisms to alter semen quality. The free radical concentration is also related to other oxidative stress parameters in serum to compare local and systemic oxidative stress. At last, the free radical concentration will also be correlated to the semen analysis parameters (WHO guidelines), lifestyle factors and food intake to detect a role for lifestyle in free radical formation and semen quality.

The main study parameters will be the free radical concentration at sperm cells and serum, correlated with microbiota in seminal plasma and related to standard semen- parameters (WHO), malondialdehyde (MDA) and free thiols concentration in blood serum, lifestyle factors and food intake.

The patients are informed about the study at their intake at the Centre of Reproductive Medicine. After informed consent, patients will have to produce semen for evaluation in the context of standard care semen analysis. A sample of that ejaculate will be collected for the SIRIUS study to measure free radicals in. Next to that, blood will be drawn from the patients at the same day as the semen analysis for the free radical measurement in serum.

Free radical measurements will be performed using diamond magnetometry. Previously, diamond magnetometry was successfully used to quantify radical formation in the acrosome of boar sperm heads. This allowed quantification of radical formation locally in real time, during capacitation. This data is not published yet and is produced in the lab of Dr. Romana Schirhagl.

Semen plasma microbiota composition will be evaluated using quantitative polymerase chain reaction (qPCR) and 16S ribosomal ribonucleic acid (rRNA) sequencing methods using QIAGEN Sample and Assay Technologies.

MDA concentration in serum will be measured using Thio barbituric acid reactive substance (TBARS) assay. Free thiol concentration in serum will be measured using the Ellman technique. A questionnaire for lifestyle factors is implemented as part of standard care for the couples seeking fertility treatment. These outcomes and answers will also be used for SIRIUS.

For an indication of food intake of the subjects a food frequency questionnaire (FFQ) of Wageningen University will be used.

ELIGIBILITY:
Inclusion Criteria:

* Males of couples visiting the CRM at the UMCG between 18-55 years old.
* Planned semen-analysis as standard care.

Exclusion Criteria:

* Males who receive(d) chemo- and/or radiotherapy, use(d) testosterone suppletion and/or anabolic steroids
* Males who are azoospermic
* Males who have an abnormal SA due to genetic causes.
* Semen analysis with round cells >2x106 /ml (as marker for infection)
* Males who currently use antibiotics

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males of couples visiting the CRM of the UMCG
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Free radical concentration in seminal plasma | Within 4 hours after production of semen at baseline
  Free radical concentration (in mola) in seminal plasma from males of couples visiting the Center of Reproductive Medicine (CRM) of the University Medical Center Groningen (UMCG) is measured using Diamond magnetometry.
Determination of seminal microbiome species and their abundance in seminal plasma | Baseline
  The different species and their relative and absolute abundance in seminal microbiota is determined in seminal plasma using qPCR and 16S rRNA sequencing methods (%).
Free radical concentration in serum using Diamond magnetometry | Within 2 hours of withdrawal at baseline
  Free radical concentration (in mola) in blood serum from males of couples visiting the Center of Reproductive Medicine (CRM) of the University Medical Center Groningen (UMCG) is measured using Diamond magnetometry.
Free thiol levels in serum using the Ellman technique | Baseline
  Free thiol levels in blood serum (in umol/L) from males of couples visiting the Center of Reproductive Medicine (CRM) of the University Medical Center Groningen (UMCG) is measured using the Ellman technique.
Malondialdehyde levels in serum using the TBARS assay | Baseline
  Malondialdehyde levels blood serum (in uM) from males of couples visiting the Center of Reproductive Medicine (CRM) of the University Medical Center Groningen (UMCG) is measured using the TBARS assay.

SECONDARY OUTCOMES:
Relation between concentration of free radicals in semen and the microbiota species composition in seminal plasma | Through study completion, an average of 1 year
  To relate the concentration of free radical in seminal plasma measured in uM with Diamond magnetometry, with the incidence of microbiota (e.g. which species and their abundance) in seminal plasma measured with qPCR and 16S rRNA sequencing methods, to detect a role of microbiota in the concentration of free radicals. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between free radical concentration in seminal plasma and free radical concentration in blood serum. | Through study completion, an average of 1 year
  To relate the concentration of free radicals in seminal plasma measured with Diamond magnetometry with the concentration of free radical in blood serum measured with Diamond magnetometry (uM), to compare systemic and local oxidative stress. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between free radical concentration in seminal plasma and free thiol levels in blood serum. | Through study completion, an average of 1 year
  To relate the concentration of free radicals in seminal plasma measured with Diamond magnetometry with the concentration of free thiols in blood serum (uM) measured with the Ellman technique (1959), to compare systemic and local oxidative stress. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between free radical concentration in seminal plasma and concentration of Malondialdehyde in blood serum. | Through study completion, an average of 1 year
  To relate the concentration of free radicals in seminal plasma measured with Diamond magnetometry with the concentration of Malondialdehyde (uM) using the thiobarbituric acid reactive substance assay (TBARS; Janero 1990), to compare systemic and local oxidative stress. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (1-5) and seminal volume measured according to the WHO guidelines. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the standard semen analysis parameter volume (cc) analyzed according to the WHO guidelines. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (1-5) and sperm concentration measured according to the WHO guidelines. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the standard semen analysis parameter sperm concentration (10^6/mL) analyzed according to the WHO guidelines. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (1-5) and semen motility measured according to the WHO guidelines. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the standard semen analysis parameter sperm motility (%/total ejaculate) analyzed according to the WHO guidelines. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and lifestyle factor: smoking, collected via routinely conducted hospital questionnaires. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the smoking habit (measured in number of cigarettes/day), to detect a role for lifestyle in male infertility. Smoking habit will be collected as part of the standard care of the couples seeking fertility treatment with a questionnaire. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and lifestyle factor: BMI, collected via routinely conducted hospital questionnaires. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the lifestyle factor BMI (kg/m^2), to detect a role for lifestyle in male infertility. BMI will be collected as part of the standard care of the couples seeking fertility treatment with a questionnaire. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and lifestyle factor: alcohol use, collected via routinely conducted hospital questionnaires. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the alcohol use (measured in units alcohol/week), to detect a role for lifestyle in male infertility. Alcohol use will be collected as part of the standard care of the couples seeking fertility treatment with a questionnaire. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and medication use collected via routinely conducted hospital questionnaires. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to medication use (measured in daily dose in mg, ml or units), to detect an influence of medication use in male infertility. Medication list will be collected as part of the standard care of the couples seeking fertility treatment with a questionnaire. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and lifestyle factor: recreative drug use, collected via routinely conducted hospital questionnaires. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to recreative drug use (measured in type and amount of drugs/week), to detect a role for lifestyle in male infertility. Drug usage will be collected as part of the standard care of the couples seeking fertility treatment with a questionnaire. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and comorbidities, collected via routinely conducted hospital questionnaires. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to the comorbidities, to detect an influence of comorbidities within male infertility. Comorbidities will be collected as part of the standard care of the couples seeking fertility treatment with a questionnaire (number of cigarettes/day, number of units of alcohol/week, type and amount of drugs use per week). Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).
Relation between primary objectives (outcome 1-5) and food intake collected using the food frequency questionnaire developed by Wageningen University. | Through study completion, an average of 1 year
  To relate the primary objectives (outcome 1-5) to food intake to detect a role for diet in male infertility. Food intake will be collected using a food frequency questionnaire (FFQ) of the University of Wageningen where previous month is used as reference point to measure the rate of specific food groups. Statistical analysis established using SPSS (IBM Corp, Armonk, NY USA).

CONTACTS AND LOCATIONS:
Overall Officials: Astrid EP Cantineau, Principal Investigator — University Medical Centre Groningen; Centre of Reproductive Medicine
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated will be stored in a non-publicly available repository, called REDCap. This is a secure web platform for building and managing online databases and surveys. All manners of identification are also accessible by public health inspectors and monitors. REDcap is Good Clinical Practive (GCP) and General Data Protection Regulation (GDPR) compliant. After the study has ended, the database is locked. For each patient a Patient Data Report will be created including notes, discrepancies and the audit file, and will be sent to the principal investigator.
  The database, blood serum and semen plasma will be kept available for as long as 15 years. Unused material will be stored and could be used for possible follow up analysis. The sperm cells will be destroyed directly after the measurements, with a maximum retention time of 48 hours. Patients will also be asked to give consent for sharing participant-level data with other research facilities/hospitals on request.

REFERENCES:
- [Background] Kumar N, Singh AK. Trends of male factor infertility, an important cause of infertility: A review of literature. J Hum Reprod Sci. 2015 Oct-Dec;8(4):191-6. doi: 10.4103/0974-1208.170370. PMID 26752853
- [Background] Tomaiuolo R, Veneruso I, Cariati F, D'Argenio V. Microbiota and Human Reproduction: The Case of Female Infertility. High Throughput. 2020 May 3;9(2):12. doi: 10.3390/ht9020012. PMID 32375241
- [Background] Mamin HJ, Kim M, Sherwood MH, Rettner CT, Ohno K, Awschalom DD, Rugar D. Nanoscale nuclear magnetic resonance with a nitrogen-vacancy spin sensor. Science. 2013 Feb 1;339(6119):557-60. doi: 10.1126/science.1231540. PMID 23372008
- [Background] Baud D, Pattaroni C, Vulliemoz N, Castella V, Marsland BJ, Stojanov M. Sperm Microbiota and Its Impact on Semen Parameters. Front Microbiol. 2019 Feb 12;10:234. doi: 10.3389/fmicb.2019.00234. eCollection 2019. PMID 30809218
- [Background] Weng SL, Chiu CM, Lin FM, Huang WC, Liang C, Yang T, Yang TL, Liu CY, Wu WY, Chang YA, Chang TH, Huang HD. Bacterial communities in semen from men of infertile couples: metagenomic sequencing reveals relationships of seminal microbiota to semen quality. PLoS One. 2014 Oct 23;9(10):e110152. doi: 10.1371/journal.pone.0110152. eCollection 2014. PMID 25340531
- [Background] Thoma ME, McLain AC, Louis JF, King RB, Trumble AC, Sundaram R, Buck Louis GM. Prevalence of infertility in the United States as estimated by the current duration approach and a traditional constructed approach. Fertil Steril. 2013 Apr;99(5):1324-1331.e1. doi: 10.1016/j.fertnstert.2012.11.037. Epub 2013 Jan 3. PMID 23290741
- [Background] Hou D, Zhou X, Zhong X, Settles ML, Herring J, Wang L, Abdo Z, Forney LJ, Xu C. Microbiota of the seminal fluid from healthy and infertile men. Fertil Steril. 2013 Nov;100(5):1261-9. doi: 10.1016/j.fertnstert.2013.07.1991. Epub 2013 Aug 29. PMID 23993888
- [Background] Agarwal A, Rana M, Qiu E, AlBunni H, Bui AD, Henkel R. Role of oxidative stress, infection and inflammation in male infertility. Andrologia. 2018 Dec;50(11):e13126. doi: 10.1111/and.13126. PMID 30569652
- [Background] DiGuiseppi J, Fridovich I. The toxicology of molecular oxygen. Crit Rev Toxicol. 1984;12(4):315-42. doi: 10.3109/10408448409044213. PMID 6204814
- [Background] Ciobanu L, Seeber DA, Pennington CH. 3D MR microscopy with resolution 3.7 microm by 3.3 microm by 3.3 microm. J Magn Reson. 2002 Sep-Oct;158(1-2):178-82. doi: 10.1016/s1090-7807(02)00071-x. PMID 12419685
- [Background] Cooper TG, Noonan E, von Eckardstein S, Auger J, Baker HW, Behre HM, Haugen TB, Kruger T, Wang C, Mbizvo MT, Vogelsong KM. World Health Organization reference values for human semen characteristics. Hum Reprod Update. 2010 May-Jun;16(3):231-45. doi: 10.1093/humupd/dmp048. Epub 2009 Nov 24. PMID 19934213
- [Background] Farahani L, Tharakan T, Yap T, Ramsay JW, Jayasena CN, Minhas S. The semen microbiome and its impact on sperm function and male fertility: A systematic review and meta-analysis. Andrology. 2021 Jan;9(1):115-144. doi: 10.1111/andr.12886. Epub 2020 Oct 7. PMID 32794312
- [Background] Bourgonje AR, Gabriels RY, de Borst MH, Bulthuis MLC, Faber KN, van Goor H, Dijkstra G. Serum Free Thiols Are Superior to Fecal Calprotectin in Reflecting Endoscopic Disease Activity in Inflammatory Bowel Disease. Antioxidants (Basel). 2019 Sep 1;8(9):351. doi: 10.3390/antiox8090351. PMID 31480545
- [Background] Janero DR. Malondialdehyde and thiobarbituric acid-reactivity as diagnostic indices of lipid peroxidation and peroxidative tissue injury. Free Radic Biol Med. 1990;9(6):515-40. doi: 10.1016/0891-5849(90)90131-2. PMID 2079232